CLINICAL TRIAL: NCT05846802
Title: Gastroparesis Registry 4 (GpR4): Improving the Understanding of Gastroparesis and Functional Dyspepsia
Brief Title: Gastroparesis Registry 4
Acronym: GpR4
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Texas Tech University Health Sciences Center, El Paso (Other); Temple University (Other); University of Louisville (Other); Mayo Clinic (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Massachusetts General Hospital (Other); Wake Forest University (Other)
Responsible Party: Sponsor
Other Study IDs: 14-DK-GpR4; U01DK073975 (NIH); U01DK074035 (NIH); U01DK074007 (NIH); U24DK074008 (NIH); U01DK073983 (NIH); U01DK112193 (NIH); U01DK073974 (NIH); IRB00401119 (Other: JHM IRB)
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Gastroparesis; Gastroparesis Nondiabetic; Gastroparesis Due to Diabetes Mellitus Type I; Gastroparesis Due to Diabetes Mellitus Type II; Functional Disorder of Gastrointestinal Tract; Gastro-Intestinal Disorder
MeSH Terms: conditions — Gastroparesis; Gastrointestinal Diseases; Digestive System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 20 mL of fasting blood collected and will be separated into plasma and serum and divided into 0.5 mL aliquots. Aliquots will be kept in a storage facility at -70 degrees C until they are shipped to the NIDDK Central Repository on dry ice for banking. The banked samples will be used for specific GpR4 research questions, GpCRC ancillary studies,and future health-related research..
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastroparesis: Gastroparesis symptoms with delayed emptying
- Functional Dyspepsia: Gastroparesis symptoms without delayed emptying

SUMMARY:
The Gastroparesis Registry 4 (GpR4) is an observational study of patients with symptoms of gastroparesis (Gp) and functional dyspepsia (FD) with either delayed or normal gastric emptying. To better understand these disorders, this registry will capture demographic, clinical, physiological, questionnaire, and patient outcome data to characterize the patients and their clinical course. Participants will complete several questionnaires, complete a nutrient drink test and have a gastric emptying study.

DETAILED DESCRIPTION:
This observational study of patients with symptoms of gastroparesis (Gp) and functional dyspepsia (FD) with either delayed or normal gastric emptying aims to assess the clinical, pathophysiological, and psychological similarities and differences between patients with Gp, FD.

The primary outcome will be the measure of symptom severity of gastroparesis and functional dyspepsia using the change in total score from the Patient Assessment of Upper Gastrointestinal Disorders Symptoms (PAGI SYM) from baseline to 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years at initial screening visit
* Symptoms of Gp and/or FD of at least 12-weeks duration with varying degrees of nausea, vomiting, early satiety, postprandial fullness, abdominal pain, abdominal burning. Thus, patients can enter the GpR4 registry primarily with abdominal pain suggesting FD-Epigastric Pain Syndrome.
* Successful completion of gastric emptying scintigraphy of solids using the 4-hour Egg Beaters® protocol (or equivalent generic liquid egg white meal) within the last 9 months
* Negative upper endoscopy or upper radiographic GI series within 5 years of registration

Exclusion Criteria:

* Use of narcotic analgesics greater than three days per week
* Presence of other conditions that could explain the patient's symptoms such as:
* Pyloric or intestinal obstruction as evidenced by EGD, UGI, or Abdominal CT
* Active inflammatory bowel disease
* Known eosinophilic gastroenteritis or eosinophilic esophagitis
* Primary neurological conditions that can cause nausea and vomiting such as increased intracranial pressure, space occupying or inflammatory/infectious lesions
* Acute or chronic renal failure (serum creatinine >3 mg/dL) and/or on hemodialysis or peritoneal dialysis
* Acute liver failure or advanced liver disease (Child's B or C; a Child-Pugh-Turcotte (CPT) score of ≥7)
* Pancreatic disorder if present on pancreatic imaging or pancreatic function testing
* Prior gastric surgery including total or subtotal (near complete) gastric resection, esophagectomy, gastrojejunostomy, gastric bypass, gastric sleeve, pyloroplasty, pyloromyotomy, or any fundoplication (Nissen, Tor)
* Any other condition, which in the opinion of the investigator, could explain the symptoms or interfere with study requirements
* Females who are pregnant. A urine pregnancy test is routinely obtained on all females immediately prior to gastric emptying procedures.
* Inability to comply with or complete the gastric emptying scintigraphy test (including allergy to eggs)
* Inability to obtain informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults over age 18, located in the United States, with symptoms of gastroparesis and/or functional dyspepsia.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Measure of symptom severity of gastroparesis and functional dyspepsia using the change in total score from the Patient Assessment of Upper Gastrointestinal Disorders Symptoms (PAGI SYM) from baseline to 48 weeks. | 48 weeks
  Change in PAGI-SYM total score from baseline to 48 weeks. The final PAGI-SYM contains 20 items grouped into 6 subscales covering:
  heartburn/regurgitation (7 items), nausea/vomiting (3 items), post-prandial fullness/early satiety (4 items), bloating (2 items), upper abdominal pain (2 items), and lower abdominal pain (2 items). A 6-point Likert response scale, ranging from 0 (none) to 5 (very severe), is used for rating the severity of each symptom item over a 2-week recall period.
  * Subscale scores vary from 0 to 5
  * Total score varies from 0 to 5
  * Lower score = better health

SECONDARY OUTCOMES:
Changes in gastric emptying, as measured by gastric emptying scintigraphy (GES) at baseline and 48 weeks | Baseline, 48 weeks
  Changes in gastric emptying, as measured by gastric emptying scintigraphy (GES) at baseline and 48 weeks.
  Normal values for gastric emptying scintigraphy have been established in earlier studies using healthy volunteers. Gastric retention of 99mTc > 60% at 2 hours and/or > 10% at 4 hours is considered evidence of delayed gastric emptying of solids.

OTHER OUTCOMES:
Presence or absence of Carnett's sign for abdominal wall pain at baseline. | Baseline
  Presence or absence Carnett's sign for abdominal wall pain at baseline. Carnett's sign is a finding on clinical examination in which (acute) abdominal pain remains unchanged or increases when the muscles of the abdominal wall are tensed. As part of the abdominal examination, the patient is asked to lift the head and shoulders from the examination table to tense the abdominal muscles. An alternative is to ask the patient to raise both legs with straight knees.
  A positive test indicates the increased likelihood that the abdominal wall and not the abdominal cavity is the source of the pain (for example, due to rectus sheath hematoma instead of appendicitis). A negative Carnett's sign is said to occur when the abdominal pain decreases when the patient is asked to lift the head; this points to an intra-abdominal cause of the pain

CONTACTS AND LOCATIONS:
Overall Officials: Jay Pasricha, MD, Principal Investigator — Mayo Clinic; Henry Parkman, MD, Principal Investigator — Temple University; David Shade, JD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (6):
- United States (6):
  - Jay Pasricha, Scottsdale, Arizona
  - University of Louisville, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Wake Forest University and Atrium Health Carolinas Medical Center, Charlotte, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Texas Tech University Health Science Center (TTUHSC), El Paso, Texas

IPD SHARING:
Plan to Share IPD: Yes
Public use complete database will be submitted to the NIDDK Data Repository
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Two years after the end of the funding period ends (2029)
Access Criteria: An investigator interested in acquiring GpR4 study data or biospecimens should contact the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Central Repository
URL: https://repository.niddk.nih.gov/home

REFERENCES:
- [Background] Parkman HP, Hasler WL, Fisher RS; American Gastroenterological Association. American Gastroenterological Association technical review on the diagnosis and treatment of gastroparesis. Gastroenterology. 2004 Nov;127(5):1592-622. doi: 10.1053/j.gastro.2004.09.055. PMID 15521026
- [Background] Camilleri M, Parkman HP, Shafi MA, Abell TL, Gerson L; American College of Gastroenterology. Clinical guideline: management of gastroparesis. Am J Gastroenterol. 2013 Jan;108(1):18-37; quiz 38. doi: 10.1038/ajg.2012.373. Epub 2012 Nov 13. PMID 23147521
- [Background] Stanghellini V, Chan FK, Hasler WL, Malagelada JR, Suzuki H, Tack J, Talley NJ. Gastroduodenal Disorders. Gastroenterology. 2016 May;150(6):1380-92. doi: 10.1053/j.gastro.2016.02.011. PMID 27147122
- [Background] Schol J, Wauters L, Dickman R, Drug V, Mulak A, Serra J, Enck P, Tack J; ESNM Gastroparesis Consensus Group. United European Gastroenterology (UEG) and European Society for Neurogastroenterology and Motility (ESNM) consensus on gastroparesis. Neurogastroenterol Motil. 2021 Aug;33(8):e14237. doi: 10.1111/nmo.14237. PMID 34399024
- [Background] Pasricha PJ, Grover M, Yates KP, Abell TL, Bernard CE, Koch KL, McCallum RW, Sarosiek I, Kuo B, Bulat R, Chen J, Shulman RJ, Lee L, Tonascia J, Miriel LA, Hamilton F, Farrugia G, Parkman HP; National Institute of Diabetes and Digestive and Kidney Diseases/National Institutes of Health Gastroparesis Clinical Research Consortium. Functional Dyspepsia and Gastroparesis in Tertiary Care are Interchangeable Syndromes With Common Clinical and Pathologic Features. Gastroenterology. 2021 May;160(6):2006-2017. doi: 10.1053/j.gastro.2021.01.230. Epub 2021 Feb 3. PMID 33548234
- [Background] Pasricha PJ, Colvin R, Yates K, Hasler WL, Abell TL, Unalp-Arida A, Nguyen L, Farrugia G, Koch KL, Parkman HP, Snape WJ, Lee L, Tonascia J, Hamilton F. Characteristics of patients with chronic unexplained nausea and vomiting and normal gastric emptying. Clin Gastroenterol Hepatol. 2011 Jul;9(7):567-76.e1-4. doi: 10.1016/j.cgh.2011.03.003. Epub 2011 Mar 11. PMID 21397732
- [Background] Makarov OV, Khashchukoeva AZ, Borisenko SA, Epeikina TN, Moiseeva NB. [Immunologic aspects of ovarian tumors]. Akush Ginekol (Mosk). 1988 Nov;(11):3-6. No abstract available. Russian. PMID 3071162
- [Background] Vijayvargiya P, Jameie-Oskooei S, Camilleri M, Chedid V, Erwin PJ, Murad MH. Association between delayed gastric emptying and upper gastrointestinal symptoms: a systematic review and meta-analysis. Gut. 2019 May;68(5):804-813. doi: 10.1136/gutjnl-2018-316405. Epub 2018 Jun 2. PMID 29860241
- [Background] Lacy BE, Crowell MD, Cangemi DJ, Lunsford TN, Simren M, Tack J. Diagnostic Evaluation of Gastric Motor and Sensory Disorders. Am J Gastroenterol. 2021 Dec 1;116(12):2345-2356. doi: 10.14309/ajg.0000000000001562. PMID 35134012
- [Background] Revicki DA, Camilleri M, Kuo B, Norton NJ, Murray L, Palsgrove A, Parkman HP. Development and content validity of a gastroparesis cardinal symptom index daily diary. Aliment Pharmacol Ther. 2009 Sep 15;30(6):670-80. doi: 10.1111/j.1365-2036.2009.04078.x. Epub 2009 Jun 25. PMID 19558608
- [Background] Yu D, Ramsey FV, Norton WF, Norton N, Schneck S, Gaetano T, Parkman HP. The Burdens, Concerns, and Quality of Life of Patients with Gastroparesis. Dig Dis Sci. 2017 Apr;62(4):879-893. doi: 10.1007/s10620-017-4456-7. Epub 2017 Jan 21. PMID 28110376
- [Background] Parkman HP, Wilson LA, Yates KP, Koch KL, Abell TL, McCallum RW, Sarosiek I, Kuo B, Malik Z, Schey R, Shulman RJ, Grover M, Farrugia G, Miriel L, Tonascia J, Hamilton F, Pasricha PJ; NIDDK/NIH Clinical Gastroparesis Consortium. Factors that contribute to the impairment of quality of life in gastroparesis. Neurogastroenterol Motil. 2021 Aug;33(8):e14087. doi: 10.1111/nmo.14087. Epub 2021 Jan 25. PMID 33493377
- [Background] Hasler WL, Wilson LA, Parkman HP, Koch KL, Abell TL, Nguyen L, Pasricha PJ, Snape WJ, McCallum RW, Sarosiek I, Farrugia G, Calles J, Lee L, Tonascia J, Unalp-Arida A, Hamilton F. Factors related to abdominal pain in gastroparesis: contrast to patients with predominant nausea and vomiting. Neurogastroenterol Motil. 2013 May;25(5):427-38, e300-1. doi: 10.1111/nmo.12091. Epub 2013 Feb 17. PMID 23414452
- [Background] Hasler WL, Wilson LA, Nguyen LA, Snape WJ, Abell TL, Koch KL, McCallum RW, Pasricha PJ, Sarosiek I, Farrugia G, Grover M, Lee LA, Miriel L, Tonascia J, Hamilton FA, Parkman HP; Gastroparesis Clinical Research Consortium. Opioid Use and Potency Are Associated With Clinical Features, Quality of Life, and Use of Resources in Patients With Gastroparesis. Clin Gastroenterol Hepatol. 2019 Jun;17(7):1285-1294.e1. doi: 10.1016/j.cgh.2018.10.013. Epub 2018 Oct 13. PMID 30326297
- [Background] Parkman HP, Wilson LA, Hasler WL, McCallum RW, Sarosiek I, Koch KL, Abell TL, Schey R, Kuo B, Snape WJ, Nguyen L, Farrugia G, Grover M, Clarke J, Miriel L, Tonascia J, Hamilton F, Pasricha PJ. Abdominal Pain in Patients with Gastroparesis: Associations with Gastroparesis Symptoms, Etiology of Gastroparesis, Gastric Emptying, Somatization, and Quality of Life. Dig Dis Sci. 2019 Aug;64(8):2242-2255. doi: 10.1007/s10620-019-05522-9. Epub 2019 Mar 9. PMID 30852767
- [Background] Glissen Brown JR, Bernstein GR, Friedenberg FK, Ehrlich AC. Chronic Abdominal Wall Pain: An Under-Recognized Diagnosis Leading to Unnecessary Testing. J Clin Gastroenterol. 2016 Nov/Dec;50(10):828-835. doi: 10.1097/MCG.0000000000000636. PMID 27548731
- [Background] Camilleri M, Chedid V, Ford AC, Haruma K, Horowitz M, Jones KL, Low PA, Park SY, Parkman HP, Stanghellini V. Gastroparesis. Nat Rev Dis Primers. 2018 Nov 1;4(1):41. doi: 10.1038/s41572-018-0038-z. PMID 30385743
- [Background] Soykan I, Sivri B, Sarosiek I, Kiernan B, McCallum RW. Demography, clinical characteristics, psychological and abuse profiles, treatment, and long-term follow-up of patients with gastroparesis. Dig Dis Sci. 1998 Nov;43(11):2398-404. doi: 10.1023/a:1026665728213. PMID 9824125
- [Background] Parkman HP, Yates K, Hasler WL, Nguyen L, Pasricha PJ, Snape WJ, Farrugia G, Koch KL, Calles J, Abell TL, McCallum RW, Lee L, Unalp-Arida A, Tonascia J, Hamilton F; National Institute of Diabetes and Digestive and Kidney Diseases Gastroparesis Clinical Research Consortium. Similarities and differences between diabetic and idiopathic gastroparesis. Clin Gastroenterol Hepatol. 2011 Dec;9(12):1056-64; quiz e133-4. doi: 10.1016/j.cgh.2011.08.013. Epub 2011 Aug 24. PMID 21871247
- [Background] Pasricha PJ, Yates KP, Nguyen L, Clarke J, Abell TL, Farrugia G, Hasler WL, Koch KL, Snape WJ, McCallum RW, Sarosiek I, Tonascia J, Miriel LA, Lee L, Hamilton F, Parkman HP. Outcomes and Factors Associated With Reduced Symptoms in Patients With Gastroparesis. Gastroenterology. 2015 Dec;149(7):1762-1774.e4. doi: 10.1053/j.gastro.2015.08.008. Epub 2015 Aug 21. PMID 26299414
- [Background] Gourcerol G, Melchior C, Wuestenberghs F, Desprez C, Prevost G, Grosjean J, Leroi AM, Tavolacci MP. Delayed gastric emptying as an independent predictor of mortality in gastroparesis. Aliment Pharmacol Ther. 2022 Apr;55(7):867-875. doi: 10.1111/apt.16827. Epub 2022 Feb 20. PMID 35187671
- [Background] Grover M, Farrugia G, Lurken MS, Bernard CE, Faussone-Pellegrini MS, Smyrk TC, Parkman HP, Abell TL, Snape WJ, Hasler WL, Unalp-Arida A, Nguyen L, Koch KL, Calles J, Lee L, Tonascia J, Hamilton FA, Pasricha PJ; NIDDK Gastroparesis Clinical Research Consortium. Cellular changes in diabetic and idiopathic gastroparesis. Gastroenterology. 2011 May;140(5):1575-85.e8. doi: 10.1053/j.gastro.2011.01.046. Epub 2011 Feb 4. PMID 21300066
- [Background] Gaddipati KV, Simonian HP, Kresge KM, Boden GH, Parkman HP. Abnormal ghrelin and pancreatic polypeptide responses in gastroparesis. Dig Dis Sci. 2006 Aug;51(8):1339-46. doi: 10.1007/s10620-005-9022-z. Epub 2006 Jul 26. PMID 16868831
- [Background] Nguyen L, Wilson LA, Miriel L, Pasricha PJ, Kuo B, Hasler WL, McCallum RW, Sarosiek I, Koch KL, Snape WJ, Farrugia G, Grover M, Clarke J, Parkman HP, Tonascia J, Hamilton F, Abell TL; NIDDK Gastroparesis Clinical Research Consortium (GpCRC). Autonomic function in gastroparesis and chronic unexplained nausea and vomiting: Relationship with etiology, gastric emptying, and symptom severity. Neurogastroenterol Motil. 2020 Aug;32(8):e13810. doi: 10.1111/nmo.13810. Epub 2020 Feb 15. PMID 32061038
- [Background] Tougas G, Eaker EY, Abell TL, Abrahamsson H, Boivin M, Chen J, Hocking MP, Quigley EM, Koch KL, Tokayer AZ, Stanghellini V, Chen Y, Huizinga JD, Ryden J, Bourgeois I, McCallum RW. Assessment of gastric emptying using a low fat meal: establishment of international control values. Am J Gastroenterol. 2000 Jun;95(6):1456-62. doi: 10.1111/j.1572-0241.2000.02076.x. PMID 10894578
- [Background] Abell TL, Camilleri M, Donohoe K, Hasler WL, Lin HC, Maurer AH, McCallum RW, Nowak T, Nusynowitz ML, Parkman HP, Shreve P, Szarka LA, Snape WJ Jr, Ziessman HA; American Neurogastroenterology and Motility Society and the Society of Nuclear Medicine. Consensus recommendations for gastric emptying scintigraphy: a joint report of the American Neurogastroenterology and Motility Society and the Society of Nuclear Medicine. Am J Gastroenterol. 2008 Mar;103(3):753-63. doi: 10.1111/j.1572-0241.2007.01636.x. Epub 2007 Nov 19. PMID 18028513
- [Background] Abell TL, Yamada G, McCallum RW, Van Natta ML, Tonascia J, Parkman HP, Koch KL, Sarosiek I, Farrugia G, Grover M, Hasler W, Nguyen L, Snape W, Kuo B, Shulman R, Hamilton FA, Pasricha PJ. Effectiveness of gastric electrical stimulation in gastroparesis: Results from a large prospectively collected database of national gastroparesis registries. Neurogastroenterol Motil. 2019 Dec;31(12):e13714. doi: 10.1111/nmo.13714. Epub 2019 Oct 4. PMID 31584238
- [Background] Sarosiek I, Van Natta M, Parkman HP, Abell T, Koch KL, Kuo B, Shulman RJ, Farrugia G, Grover M, Hamilton FA, Pasricha PJ, Yates KP, Miriel L, Wilson L, Yamada G, Tonascia J, McCallum RW; National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Gastroparesis Clinical Research Consortium (GpCRC). Effect of Domperidone Therapy on Gastroparesis Symptoms: Results of a Dynamic Cohort Study by NIDDK Gastroparesis Consortium. Clin Gastroenterol Hepatol. 2022 Mar;20(3):e452-e464. doi: 10.1016/j.cgh.2021.05.063. Epub 2021 Jun 2. PMID 34089855
- [Background] Revicki DA, Rentz AM, Dubois D, Kahrilas P, Stanghellini V, Talley NJ, Tack J. Development and validation of a patient-assessed gastroparesis symptom severity measure: the Gastroparesis Cardinal Symptom Index. Aliment Pharmacol Ther. 2003 Jul 1;18(1):141-50. doi: 10.1046/j.1365-2036.2003.01612.x. PMID 12848636
- [Background] Fraser A, Delaney BC, Ford AC, Qume M, Moayyedi P. The Short-Form Leeds Dyspepsia Questionnaire validation study. Aliment Pharmacol Ther. 2007 Feb 15;25(4):477-86. doi: 10.1111/j.1365-2036.2006.03233.x. PMID 17270004
- [Background] Orthey P, Yu D, Van Natta ML, Ramsey FV, Diaz JR, Bennett PA, Iagaru AH, Fragomeni RS, McCallum RW, Sarosiek I, Hasler WL, Farrugia G, Grover M, Koch KL, Nguyen L, Snape WJ, Abell TL, Pasricha PJ, Tonascia J, Hamilton F, Parkman HP, Maurer AH; NIH Gastroparesis Consortium. Intragastric Meal Distribution During Gastric Emptying Scintigraphy for Assessment of Fundic Accommodation: Correlation with Symptoms of Gastroparesis. J Nucl Med. 2018 Apr;59(4):691-697. doi: 10.2967/jnumed.117.197053. Epub 2017 Sep 28. PMID 28970332
- [Background] Scarpellini E, Van den Houte K, Schol J, Huang IH, Colomier E, Carbone F, Tack J. Nutrient Drinking Test as Biomarker in Functional Dyspepsia. Am J Gastroenterol. 2021 Jul 1;116(7):1387-1395. doi: 10.14309/ajg.0000000000001242. PMID 33941747
- [Background] Koch KL, Hasler WL, Van Natta M, Calles-Escandon J, Grover M, Pasricha PJ, Snape WJ, Parkman HP, Abell TL, McCallum RW, Nguyen LA, Sarosiek I, Farrugia G, Tonascia J, Lee L, Miriel L, Hamilton F; NIDDK Gastroparesis Clinical Research Consortium. Satiety testing in diabetic gastroparesis: Effects of insulin pump therapy with continuous glucose monitoring on upper gastrointestinal symptoms and gastric myoelectrical activity. Neurogastroenterol Motil. 2020 Jan;32(1):e13720. doi: 10.1111/nmo.13720. Epub 2019 Oct 1. PMID 31574209
- [Background] Parkman HP, Jones MP. Tests of gastric neuromuscular function. Gastroenterology. 2009 May;136(5):1526-43. doi: 10.1053/j.gastro.2009.02.039. Epub 2009 Mar 16. PMID 19293005
- [Background] Chial HJ, Camilleri C, Delgado-Aros S, Burton D, Thomforde G, Ferber I, Camilleri M. A nutrient drink test to assess maximum tolerated volume and postprandial symptoms: effects of gender, body mass index and age in health. Neurogastroenterol Motil. 2002 Jun;14(3):249-53. doi: 10.1046/j.1365-2982.2002.00326.x. PMID 12061909
- [Background] Delgado-Aros S, Cremonini F, Castillo JE, Chial HJ, Burton DD, Ferber I, Camilleri M. Independent influences of body mass and gastric volumes on satiation in humans. Gastroenterology. 2004 Feb;126(2):432-40. doi: 10.1053/j.gastro.2003.11.007. PMID 14762780
- [Background] Mottalib A, Abrahamson MJ, Pober DM, Polak R, Eldib AH, Tomah S, Ashrafzadeh S, Hamdy O. Effect of diabetes-specific nutrition formulas on satiety and hunger hormones in patients with type 2 diabetes. Nutr Diabetes. 2019 Sep 24;9(1):26. doi: 10.1038/s41387-019-0093-x. PMID 31551412
- [Background] Phillips AE, Faghih M, Kuhlmann L, Larsen IM, Drewes AM, Singh VK, Yadav D, Olesen SS; Pancreatic Quantitative Sensory Testing (P-QST) Consortium. A clinically feasible method for the assessment and characterization of pain in patients with chronic pancreatitis. Pancreatology. 2020 Jan;20(1):25-34. doi: 10.1016/j.pan.2019.11.007. Epub 2019 Nov 20. PMID 31787527
- [Background] Sletten DM, Suarez GA, Low PA, Mandrekar J, Singer W. COMPASS 31: a refined and abbreviated Composite Autonomic Symptom Score. Mayo Clin Proc. 2012 Dec;87(12):1196-201. doi: 10.1016/j.mayocp.2012.10.013. PMID 23218087
- [Background] Song J, Bhuta R, Baig K, Parkman HP, Malik Z. COVID-19 infection manifesting as a severe gastroparesis flare: A case report. Medicine (Baltimore). 2021 Apr 9;100(14):e25467. doi: 10.1097/MD.0000000000025467. PMID 33832159
- [Background] Palsson OS, Whitehead WE, van Tilburg MA, Chang L, Chey W, Crowell MD, Keefer L, Lembo AJ, Parkman HP, Rao SS, Sperber A, Spiegel B, Tack J, Vanner S, Walker LS, Whorwell P, Yang Y. Rome IV Diagnostic Questionnaires and Tables for Investigators and Clinicians. Gastroenterology. 2016 Feb 13:S0016-5085(16)00180-3. doi: 10.1053/j.gastro.2016.02.014. Online ahead of print. PMID 27144634
- [Background] Talley NJ, Verlinden M, Jones M. Quality of life in functional dyspepsia: responsiveness of the Nepean Dyspepsia Index and development of a new 10-item short form. Aliment Pharmacol Ther. 2001 Feb;15(2):207-16. doi: 10.1046/j.1365-2036.2001.00900.x. PMID 11148439
- [Background] de la Loge C, Trudeau E, Marquis P, Kahrilas P, Stanghellini V, Talley NJ, Tack J, Revicki DA, Rentz AM, Dubois D. Cross-cultural development and validation of a patient self-administered questionnaire to assess quality of life in upper gastrointestinal disorders: the PAGI-QOL. Qual Life Res. 2004 Dec;13(10):1751-62. doi: 10.1007/s11136-004-8751-3. PMID 15651545
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-15: validity of a new measure for evaluating the severity of somatic symptoms. Psychosom Med. 2002 Mar-Apr;64(2):258-66. doi: 10.1097/00006842-200203000-00008. PMID 11914441
- [Background] Taylor F, Higgins S, Carson RT, Eremenco S, Foley C, Lacy BE, Parkman HP, Reasner DS, Shields AL, Tack J, Talley NJ; Patient-Reported Outcome Consortium's Functional Dyspepsia Working Group. Development of a Symptom-Focused Patient-Reported Outcome Measure for Functional Dyspepsia: The Functional Dyspepsia Symptom Diary (FDSD). Am J Gastroenterol. 2018 Jan;113(1):39-48. doi: 10.1038/ajg.2017.265. Epub 2017 Sep 19. PMID 28925989
- [Background] Hasler WL, Parkman HP, Wilson LA, Pasricha PJ, Koch KL, Abell TL, Snape WJ, Farrugia G, Lee L, Tonascia J, Unalp-Arida A, Hamilton F; NIDDK Gastroparesis Clinical Research Consortium. Psychological dysfunction is associated with symptom severity but not disease etiology or degree of gastric retention in patients with gastroparesis. Am J Gastroenterol. 2010 Nov;105(11):2357-67. doi: 10.1038/ajg.2010.253. Epub 2010 Jun 29. PMID 20588262
- [Background] DiBaise JK, Patel N, Noelting J, Dueck AC, Roarke M, Crowell MD. The relationship among gastroparetic symptoms, quality of life, and gastric emptying in patients referred for gastric emptying testing. Neurogastroenterol Motil. 2016 Feb;28(2):234-42. doi: 10.1111/nmo.12718. Epub 2015 Nov 7. PMID 26547484
- [Background] Parkman HP, Hallinan EK, Hasler WL, Farrugia G, Koch KL, Calles J, Snape WJ, Abell TL, Sarosiek I, McCallum RW, Nguyen L, Pasricha PJ, Clarke J, Miriel L, Lee L, Tonascia J, Hamilton F; NIDDK Gastroparesis Clinical Research Consortium (GpCRC). Nausea and vomiting in gastroparesis: similarities and differences in idiopathic and diabetic gastroparesis. Neurogastroenterol Motil. 2016 Dec;28(12):1902-1914. doi: 10.1111/nmo.12893. Epub 2016 Jun 27. PMID 27350152
- [Background] Hasler WL, Wilson LA, Parkman HP, Nguyen L, Abell TL, Koch KL, Pasricha PJ, Snape WJ, Farrugia G, Lee L, Tonascia J, Unalp-Arida A, Hamilton F; NIDDK Gastroparesis Clinical Research Consortium (GpCRC). Bloating in gastroparesis: severity, impact, and associated factors. Am J Gastroenterol. 2011 Aug;106(8):1492-502. doi: 10.1038/ajg.2011.81. Epub 2011 Apr 12. PMID 21483459
- [Background] Abell TL, Bernstein RK, Cutts T, Farrugia G, Forster J, Hasler WL, McCallum RW, Olden KW, Parkman HP, Parrish CR, Pasricha PJ, Prather CM, Soffer EE, Twillman R, Vinik AI. Treatment of gastroparesis: a multidisciplinary clinical review. Neurogastroenterol Motil. 2006 Apr;18(4):263-83. doi: 10.1111/j.1365-2982.2006.00760.x. PMID 16553582
- [Background] Pasricha PJ, Camilleri M, Hasler WL, Parkman HP. White Paper AGA: Gastroparesis: Clinical and Regulatory Insights for Clinical Trials. Clin Gastroenterol Hepatol. 2017 Aug;15(8):1184-1190. doi: 10.1016/j.cgh.2017.04.011. Epub 2017 Apr 12. PMID 28410896
- [Background] Parkman HP, Yates KP, Hasler WL, Nguyan L, Pasricha PJ, Snape WJ, Farrugia G, Calles J, Koch KL, Abell TL, McCallum RW, Petito D, Parrish CR, Duffy F, Lee L, Unalp-Arida A, Tonascia J, Hamilton F; NIDDK Gastroparesis Clinical Research Consortium. Dietary intake and nutritional deficiencies in patients with diabetic or idiopathic gastroparesis. Gastroenterology. 2011 Aug;141(2):486-98, 498.e1-7. doi: 10.1053/j.gastro.2011.04.045. Epub 2011 Apr 28. PMID 21684286
- [Background] Parkman HP, Yates K, Hasler WL, Nguyen L, Pasricha PJ, Snape WJ, Farrugia G, Koch KL, Abell TL, McCallum RW, Lee L, Unalp-Arida A, Tonascia J, Hamilton F; National Institute of Diabetes and Digestive and Kidney Diseases Gastroparesis Clinical Research Consortium. Clinical features of idiopathic gastroparesis vary with sex, body mass, symptom onset, delay in gastric emptying, and gastroparesis severity. Gastroenterology. 2011 Jan;140(1):101-15. doi: 10.1053/j.gastro.2010.10.015. Epub 2010 Oct 20. PMID 20965184